CLINICAL TRIAL: NCT05995431
Title: Impact of Bruxism in the Outcome of Subgingival Instrumentation for the Management of Stage 2 and Stage 3 Periodontitis: A Comparative Interventional Study.
Brief Title: Impact of Bruxism in the Outcome of Subgingival Instrumentation for the Management of Stage 2 and Stage 3 Periodontitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIYANKAPERIO2023
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Bruxism
MeSH Terms: conditions — Periodontitis; Bruxism | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERIODONTITIS STAGE 2 AND STAGE 3 WITH BRUXISM (Experimental): All the participants will undergo scaling and root planing
  Interventions: Procedure: scaling and root planing
- AGE MATCHED PATIENTS WITH STAGE 2 AND STAGE 3 PERIODONTITIS WITHOUT BRUXISM (Active Comparator): All the participants will undergo subgingival instrumentation
  Interventions: Procedure: Subgingival instrumentation

INTERVENTIONS:
Procedure: scaling and root planing — All the participants will undergo scaling and root planing
  Other Names: SRP
  Arms: PERIODONTITIS STAGE 2 AND STAGE 3 WITH BRUXISM
Procedure: Subgingival instrumentation — All the participants will undergo subgingival instrumentation
  Arms: AGE MATCHED PATIENTS WITH STAGE 2 AND STAGE 3 PERIODONTITIS WITHOUT BRUXISM

SUMMARY:
Bruxism is a multifaceted phenomenon that has been associated with several factors mediated by the central nervous system3. Bruxism is an umbrella term grouping different motor phenomenon. 'Bruxism is a repetitive jaw-muscle activity characterized by clenching or grinding of the teeth and/or by bracing or thrusting of the mandible. Bruxism has two distinct circadian manifestations: it can occur during sleep (indicated as sleep bruxism) or during wakefulness (indicated as awake bruxism5.

Sleep bruxism is considered to be a putative exacerbating factor, rather than a causative factor of periodontal disease and night-guards have been used as a counter measure. Since the periodontium in sleep bruxism patients suffers from excessive occlusal force for long periods of time during sleep, the function of the periodontium in such patients may differ from that in patients without sleep bruxism. Awake bruxism is defined as masticatory muscle activity during wakefulness that is characterized by repetitive or sustained tooth contact and by bracing or thrusting of the mandible.Given the potential impact of abnormal forces on the periodontium, understanding the relationship between bruxism and periodontal disease is crucial for the prevention and management of these conditions. This study aims to explore the mechanisms by which bruxism affects the periodontium and to assess the impact of bruxism in the outcome of subgingival instrumentation for the management of Stage 2 and Stage 3 periodontitis.

DETAILED DESCRIPTION:
AIM : To study the impact of bruxism in the outcome of subgingival instrumentation for the management of Stage 2 and Stage 3 periodontitis.

OBJECTIVES:

To assess the association of bruxism with periodontitis. STUDY DESIGN: An interventional study will be conducted in the Department of Periodontics and Oral implantology PGIDS, Rohtak.

STUDY SETTING: Hospital based study- patients diagnosed with Stage 2 and Stage 3 Periodontitis associated with bruxism will be recruited in study from OPD.

TIME FRAME: 12-14 months

Sociodemographic variables:

Sociodemographic data comprises of :

1. Gender
2. Age
3. Educational level,
4. Occupation status (student, employed, unemployed or retired), 5 Marital status (single, married, divorced or widowed),

6. Average family monthly income.

POPULATION:

Systemically healthy patients with generalized periodontitis : stage 2 and stage 3 of age group of 30-50 years will be recruited in the study from OPD of Periodontology. Recruitment of the patients for the study will be based on eligibility criteria after obtaining informed and written consent.

SAMPLE SIZE:

Sample size determination was done by using G power software. Taking alpha= 0.5 and power of 90% , minimum 23 patients in each group are required to detect a clinically relevant change of 1mm in clinical attachment level with standard deviation of 1mm between both the groups. Hence a total of 58 patients (29 in each group) will be included in the study expecting a 25% drop out rate.

METHOD:

Patients fulfilling the eligibility criteria will be enrolled in the study after obtaining the informed consent. Periodontal parameters will be assessed which include clinical attachment level (CAL), periodontal pocket depth (PPD), bleeding on probing (BOP), Gingival index (GI),Tooth mobility.

SAMPLE SIZE:

Sample size determination was done by using G power software. Taking alpha= 0.5 and power of 90% , minimum 23 patients in each group are required to detect a clinically relevant change of 1mm in clinical attachment level with standard deviation of 1mm between both the groups. Hence a total of 58 patients (29 in each group) will be included in the study expecting a 25% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

TEST GROUP

* Systemically healthy patients
* Patient having stage 2 or stage 3 periodontitis with bruxism Age between 30-50 years
* Minimum 20 teeth present in oral cavity

CONTROL GROUP

* Systemically healthy patients
* Patient having stage 2 or stage 3 periodontitis without bruxism
* Age between 30-50 years
* Minimum 20 teeth present in oral cavity

Exclusion Criteria:

* History of systemic disease such as diabetes or autoimmune disease
* History of drugs having the potential impact on periodontal status like phenytoin, cyclosporin, calcium-channel blockers or antidepressant drugs
* Pregnant or lactating females

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) | BASELINE,2 MONTHS ,3 MONTHS,6 MONTHS
  CLINICAL ATTACHMENT LEVEL(CAL) Clinical Attachment Level will be measured as a distance betweenfrom the base of the clinicalpocket and the cemencemento-enamel junction (CEJ).Measurements will be made atsites 6 of involved tooth- mesio-buccal, mid-buccal, dismdistobuccal, mesio-lingual, mid-lingual, disto-lingual using UNC-15 probe. Measurements will be rounded to the nearest whole millimetre.
Bleeding on probing (BOP) | BASELINE,2 MONTHS,3 MONTHS 6 MONTHS
  BLEEDING ON PROBING (BOP) BOP will recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as
  % sites with bleeding on probing.
Pocket Probing Depth (PPD) | BASELINE, 2 MONTHS, 3MONTHS, 6 MONTHS
  PROBING POCKET DEPTH (PD):Probing pocket depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP- UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of involved tooth - mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual. Measurements will be rounded to the nearest whole millimetre.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Chandela, BDS, Principal Investigator — PT BD SHARMA UHSR, HARYANA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No